CLINICAL TRIAL: NCT05818215
Title: The Impact of the Qatar 2022 FIFA World Cup During Winter Epidemics on Paediatric Emergency Department Use and Misuse Patterns: a Multicentre, Retrospective, Population-based Study
Brief Title: Impact of the Qatar 2022 FIFA World Cup on PED Use and Misuse Patterns
Status: Completed | Type: Observational
Sponsor: Pediatric Clinical Research Platform (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Johan Siebert, MD, Principal Investigator, Pediatric Clinical Research Platform
Other Study IDs: FIFA World Cup Qatar 2022
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Emergencies; Epidemic Disease; Pediatric ALL; Electronic Medical Record
Keywords: Pediatric Emergency Medicine; Emergency Service Hospital; Pediatrics; Epidemics; Respiratory Syncytial Viruses; Influenza, Human; SARS-CoV-2; Sports
MeSH Terms: conditions — Emergencies; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Data from electronic medical records of all patients under 16 years of age with medical, surgical and traumatology emergencies attending the paediatric emergency departments during the study period
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention — NO intervention

SUMMARY:
A retrospective cohort study to explore the impact of the FIFA World Cup 2022 Qatar on paediatric emergency department attendance at two tertiary centres during unprecedent winter viral epidemics.

DETAILED DESCRIPTION:
Earlier studies have reported contradictory relationship between major sporting events and paediatric emergency department attendance. None were conducted during an epidemic surge. The FIFA football World Cup 2022 was held for the first time in its history during the winter period in the northern hemisphere during unprecedented cumulative waves of respiratory syncitial virus (RSV), influenza and severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) epidemics.

This study aims to measure the impact of such a global major sporting events on the pattern of paediatric emergency department use and hospital admissions during a peak epidemic season in 2 tertiary hospitals. The study hypothesis was that major sporting events, even during an epidemic peak, can reduce the number of paediatric emergency department visits compared with periods without a sporting event. Major sporting events could serve as a model for identifying human behaviours and patterns leading to paediatric emergency department misuse, in order to develop public health interventions to better rationalise health-seeking behaviours.

ELIGIBILITY:
Inclusion Criteria:

* all patients

Exclusion Criteria:

* none

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients under 16 years of age with medical, surgical and traumatology emergencies attending each pediatric emergency department during the study period will be included. This also includes transfer cases from other hospitals, as well as those who leave prematurely without being seen.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
PED visits | Institutional electronic medical records analysed retrospectively from October 1st, 2022 to December 31, 2022
  Retrospective analysis of number of PED visits (counts).

SECONDARY OUTCOMES:
Triage acuity score | Institutional electronic medical records analysed retrospectively from October 1st, 2022 to December 31, 2022
  Retrospective analysis of number of PED visits (counts) by triage acuity score (coded using the 5-level Canadian Triage and Acuity Scale (from level 1 [resuscitation] to level 5 [nonurgent]).
Chief complaint | Institutional electronic medical records analysed retrospectively from October 1st, 2022 to December 31, 2022
  Retrospective analysis of number of PED visits (counts) by chief complaints.
Main diagnosis | Institutional electronic medical records analysed retrospectively from October 1st, 2022 to December 31, 2022
  Retrospective analysis of number of PED visits (counts) by main diagnosis (coded using the International Classification of Primary Care, 2nd edition [ICPC-2], and International Statistical Classification of Diseases and Related Health Problems, 10th revision [ICD-10-GM]).
Audience | Analysed retrospectively from October 1st, 2022 to December 31, 2022
  Daily television and online media audience collected by the independent, multi-platform Swiss national foundation for media research (Mediapulse AG, Bern, Switzerland).
RSV incidence | Analysed retrospectively from October 1st, 2022 to December 31, 2022
  RSV-incidence estimates among children will be obtained from the anonymised Swiss RSV EpiCH multicentre database. RSV testing uses reverse-transcription polymerase chain reaction or rapid antigen test at the point of care.
Influenza incidence | Analysed retrospectively from October 1st, 2022 to December 31, 2022
  Influenza-incidence among children visiting the PED during the study period will be obtained from the institutional electronic medical records. RSV testing on nasopharyngeal swabs uses reverse-transcription polymerase chain reaction at the point of care.
SARS-CoV-2 incidence | Analysed retrospectively from October 1st, 2022 to December 31, 2022
  SARS-CoV-2-incidence among children visiting the PED during the study period will be obtained from the institutional electronic medical records. SARS-CoV-2 testing on nasopharyngeal swabs uses reverse-transcription polymerase chain reaction at the point of care.

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Siebert, MD, Study Director — Geneva Children's Hospital, Geneva University Hospitals, Geneva, Switzerland
Locations (1):
- Geneva Children's Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be deidentified and the study investigators will house the data locally on secured servers at the Geneva University Hospitals. The datasets used or analysed during the current trial will be available from the corresponding author upon reasonable request. Only deidentified/anonymised data will be shared.
Time Frame: Available from 6 month to 5 years after trial publication.
Access Criteria: * Data will be made available from the corresponding author upon approval of a proposal and with a signed data access agreement.
  * Data will be made available for a specified research purpose.
  * The request proposal must include a statistician.